CLINICAL TRIAL: NCT04910490
Title: A Descriptive Research on the Effect of Primary Brainstem Hemorrhage Stereotactic Aspiration Based on 'Zhe-er Classification'
Brief Title: Stereotactic Aspiration for Primary Brainstem Hemorrhage Based on 'Zhe-er Classification'
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-908
Record Dates: First submitted 2021-05-31; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Primary Brainstem Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients received stereotaxic aspiration: No new/additional patients will be enrolled within this project. Only retrospective data will be collected on survival time and life quality
  Interventions: Other: No interventions - retrospective data collection
- Patients received conservative therapy: No new/additional patients will be enrolled within this project. Only retrospective data will be collected on survival time and life quality
  Interventions: Other: No interventions - retrospective data collection

INTERVENTIONS:
Other: No interventions - retrospective data collection — No new/additional patients will be enrolled within this project.

SUMMARY:
The purpose of this study is to determine the benefit of stereotaxic aspiration for patients with primary brainstem hemorrhage with the guidance of 'Zhe-er Classification'

DETAILED DESCRIPTION:
This is a retrospective study aiming to analyze the clinical record of patients from March 2014 to October 2020. This study is indicated for primary brainstem hemorrhage.

ELIGIBILITY:
no new patients will be enrolled within this project

Inclusion Criteria:

* Patients undergoing a stereotaxic aspiration or conservative therapy from 3/2014 to 10/2020 in 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China

Exclusion Criteria:

* patients with secondary brainstem hemorrhage due to blood vessel malformation, trauma, or malignancies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with primary brainstem hemorrhage who receive stereotaxic aspiration or conservative therapy from 3/2014 to 10/2020 in 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival events | 1 year after hemorrhage
  Survival events include death, deterioration/recovery of nervous function

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Zhang, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Jianmin Zhang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou J, Wang R, Mao J, Gu Y, Shao A, Liu F, Zhang J. Prognostic models for survival and consciousness in patients with primary brainstem hemorrhage. Front Neurol. 2023 Feb 23;14:1126585. doi: 10.3389/fneur.2023.1126585. eCollection 2023. PMID 36908614